CLINICAL TRIAL: NCT01387256
Title: Comparing Two Regimens for Medical Abortion: Mifepristone + Misoprostol Versus Misoprostol Alone-3 Hour Intervals
Brief Title: Comparing Two Regimens for Medical Abortion: Mifepristone + Misoprostol Versus Misoprostol Alone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Dr Beverly Winikoff, Gynuity Health Projects
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1.2.1
Record Dates: First submitted 2011-05-02; First posted 2011-07-04 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Complete Abortion
Keywords: abortion; mifepristone; misoprostol; with gestations > 63 days LMP

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- mifepristone+misoprostol (Other): 200 mg mifepristone + 800 mcg buccal misoprostol
  Interventions: Drug: medical abortion
- buccal misoprostol (Experimental): 2 doses of 800 mcg buccal misoprostol
  Interventions: Drug: medical abortion

INTERVENTIONS:
Drug: medical abortion — pregnancy termination with drugs

SUMMARY:
This double blinded, placebo-controlled randomized trial will compare the safety, efficacy and acceptability of two medical abortion regimens up to 63 days since last Menstrual Period (LMP) in Tunisia and Vietnam. The first regimen will include a 200 mg oral dose of mifepristone followed by 800 mcg buccal misoprostol. The second regimen will include two 800 mcg doses of buccal misoprostol three hours apart. All drugs are administered AT home by the participant.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age < 63 days since LMP, confirmed by ultrasound or clinical assessment.
* General good health including absence of conditions which contraindicate the use of mifepristone and misoprostol for pregnancy termination.
* Agrees to return for follow-up visit and willing to provide an address and/or telephone number for purposes of follow-up.
* Able to consent to study participation.

Exclusion Criteria:

* Gestational age > 63 days LMP
* Confirmed or suspected ectopic or molar pregnancy
* Contraindications to medical abortion including intra-uterine device (IUD) in place (must be removed before procedure), chronic adrenal failure, concurrent long-term corticosteroid therapy, history of allergy to mifepristone, misoprostol or prostaglandin, hemorrhagic disorders or concurrent anticoagulant therapy, inherited porphyries.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2009-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Number of women with a complete abortion using study drug alone without recourse to surgical intervention | one week from initial treatment
  Number of participants with a complete abortion after treatment without recourse to surgical intervention as a measure of efficacy of the study regimens

SECONDARY OUTCOMES:
Number of women who indicate that the side effects of buccal misoprostol, administered either alone or in combination with mifepristone, is acceptable in Tunisia and Vietnam | one week from initial treatment
  Proportion of women who report the side effects after their treatment to be acceptable as a measure of acceptability with the buccal misoprostol route (with and without mifepristone)
Evaluate whether women administering buccal misoprostol have a complete abortion with study drug and experience any adverse events, at a rate that is similar to other routes of misoprostol administration | one week from initial treatment
  To assess the rate of complete uterine evacuation with study drugs alone and rate of any adverse events among participants after use of buccal misoprostol (alone or with mifepristone)as a measure of its utility in early medical abortion compared to other regimens
Measuring the proportion of women who report their medical abortion procedure to be acceptable in Tunisia and Vietnam | one week from initial treatment
  Proportion of participants reporting that they found the medical abortion regimen assigned to them to be acceptable
Determining whether women can take both the mifepristone and misoprostol at home on their own by assessing protocol compliance | one week from initial treatment
  Proportion of women who report taking mifepristone and misoprostol at home on their own as instructed as a measure of compliance and feasibility of a protocol with at home administration of study drugs

CONTACTS AND LOCATIONS:
Locations (2):
- La Rabta Maternity Hospital, Tunis, Tunisia
- Hung Vuong Hospital, Ho Chi Minh City, Vietnam